CLINICAL TRIAL: NCT04974853
Title: Cholesterol Lowering Effect of Cardio-Complement, an Ayurveda Formulation: Feasibility Study on Patients With Mild-to-moderate Hypercholesterolemia
Brief Title: Cholesterol Lowering Effect of Cardio-Complement, an Ayurveda Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/Aaro/21-11
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-06

CONDITIONS: Hypercholesterolemia
Keywords: Ayurveda; Cholesterol; Cardiovascular Diseases; Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda Formulation (Experimental): Patients with hypercholesterolemia treated with Ayurveda formulation, Cardio-Complement
  Interventions: Combination Product: Cardio-complement

INTERVENTIONS:
Combination Product: Cardio-complement — Ayurvedic combination of Terminalia Arjuna, Withania Sominifera, Garcinia Cambogia and piperine (as bioenhancer) in pre-specified dosage.

SUMMARY:
The aim of this feasibility study was to assess the lipid-lowering effects and safety of a Ayurveda formulation containing Terminalia Arjuna, Withania Sominifera, Garcinia Cambogia and piperine (as bioenhancer)

DETAILED DESCRIPTION:
The COVID-19 related lockdowns severely affected the healthcare in India, specially in second wave of COVID-19. This research presents the applicability of Ayurveda formulation to analyze the impact on lipid profile during the lockdown.

Patients with hyperlipidemia who referred to Gyansanjeevani were recruited. All participants were enrolled in the study after a complete physical examination and medical history remotely over the virtual secure platform.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* BMI between 18.5 and 40 kg/m2
* Total Cholesterol >180 mg/dl
* No clinically significant medical history
* Willing to participate to the study by complying with the protocol
* Able to provide written informed consent

Exclusion Criteria:

* Metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder,
* Severe chronic disease
* History of ischemic cardiovascular event,
* Uncontrolled hypertension
* Under treatment or dietary supplement which could affect study parameter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Reduction of LDL-cholesterol | Change from baseline to 2 weeks

SECONDARY OUTCOMES:
Reduction of total cholesterol | Changes from baseline to 2 weeks
Increase of HDL cholesterol | Change from baseline to 2 weeks
Reduction of Triglycerides | Change from baseline to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prashanna T Chockalingam, Principal Investigator — NMP Medical Research Institute, India; Abhijit Venu, Study Chair — Aarogyam UK; Skanthesh Lakshmanan, Study Director — NMP Medical Research Institute, India
Locations (1):
- Gyansanjeevani, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided